CLINICAL TRIAL: NCT03138668
Title: The Influence of Different Doses of Local Anesthetic on the Distribution of Anesthesia of the Lateral Femoral Cutaneous Nerve - a Randomized, Blinded, Paired Study of Healthy Individuals
Brief Title: Cutaneous Anesthesia of the Lateral Femoral Cutaneous Nerve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SM2-KHT-2016; 2016-004936-39 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-03

CONDITIONS: Nerve Block; Anesthesia, Local; Pain, Postoperative; Anatomical Distribution; Nervus Cutaneous Femoris Lateralis; Lateral Femoral Cutaneous Nerve
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose Ropivacaine (Experimental): Perineural injection of 8 ml of Ropivacaine 0.75% at the lateral femoral cutaneous nerve
  Interventions: Drug: Ropivacaine Injection
- High dose Ropivacaine (Experimental): Perineural injection of 16 ml of Ropivacaine 0.75% at the lateral femoral cutaneous nerve.
  Interventions: Drug: Ropivacaine Injection

INTERVENTIONS:
Drug: Ropivacaine Injection — All 20 study participants will receive both treatment "Low dose Ropivacaine" and "High dose Ropivacaine" in form of a nerve block injection around the lateral femoral cutaneous nerve. Treatment "Low dose Ropivacaine" and "High dose Ropivacaine" will be randomized to be given in either right or left lower extremity. If the participant is randomized to receive treatment "Low dose Ropivacaine" in the right lower extremity, treatment "High dose Ropivacaine" will be given in the left lower extremity, and vice versa. Each participant will thus constitute as their own control.
  Other Names: 8 ml Ropivacaine 0.75%
  Arms: Low dose Ropivacaine
Drug: Ropivacaine Injection — All 20 study participants will receive both treatment "Low dose Ropivacaine" and "High dose Ropivacaine" in form of a nerve block injection around the lateral femoral cutaneous nerve. Treatment "Low dose Ropivacaine" and "High dose Ropivacaine" will be randomized to be given in either right or left lower extremity. If the participant is randomized to receive treatment "Low dose Ropivacaine" in the right lower extremity, treatment "High dose Ropivacaine" will be given in the left lower extremity, and vice versa. Each participant will thus constitute as their own control.
  Other Names: 16 ml Ropivacaine 0.75%
  Arms: High dose Ropivacaine

SUMMARY:
The purpose of this study is to investigate and describe the anatomical differences in distribution of the blocked area following a perineural LFCN (Lateral Femoris Cutaneous Nerve) block with either 8 ml or 16 ml of Ropivacaine, in relation to incision lines used in THA (Total Hip Arthroplasty). Furthermore, we examine any loss of motor function in Musculus Quadriceps due to posible involvement of the Femoral Nerve. This trial will be conducted in healthy volunteers, as a blinded, randomized, paired trial.

DETAILED DESCRIPTION:
Background:

Total hip arthroplasties may be associated with moderate to intense postoperative pain. It is essential that pain treatment, besides being analgesic, has a minimum of side effects, especially those opioid-related, in order to achieve low morbidity, high patient satisfaction and to encourage the functional rehabilitation.

Currently, there is no "gold standard" for pain treatment after THA, and there exists a large variety of treatment options. Some patients who have undergone THA, can be difficult to sufficiently treat with conventional analgesics without reaching additional morphine doses where side effects are unacceptable. It is therefore important to explore other treatment options, including nerve blockade.

Nerve blocks have previously been used after THA operations, but have been hampered by the fact, that the nerve blocks have an effect on the motorial nerve, inhibiting early mobilization and possibly increasing tendencies to fall when mobilized. The Lateral Femoral Cutaneous Nerve (LFCN) is purely sensorial and can therefore relieve the patient of pain without influencing the early mobilization.

In two previous trials, the investigators have studied the effect of LFCN blocks in pain treatment after THA. In the recent study, the LFCN block was applied in patients after THA, who still had visual analogue scale (VAS) mobilization pain > 40 mm when lifting their leg stretched. The LFCN block alleviated significantly the average pain at group level. Meanwhile 42% of patients in the study had no or limited effect of the block. The reason for this may be due to the fact, that LFCN block does not cover all types of pain after THA, but also the fact, that the nerve innervation area has individual differences in the anatomical distribution. We are currently investigating this matter in another study.

LFCN arise from the lumbar plexus, L1-L3. It progresses profound to m. psoas major and over m. iliacus towards the anterior superior iliac spine (ASIS). LFCN perforates the inguinal ligament in varying distance from the ASIS. Afterwards it makes a roughly 90 degrees lateral turn, divides into 3-5 branches and innervates skin lying on the lateral, proximal part of the leg. LFCN is found to have multiple anatomical variations therefore it is described to innervate both the lateral, as well as the anterior, parts of the thigh.

A single study has described LFCN as being placed in it's own canal created by a splitting of the Iliac Fascia creating a lumen in which the nerve lies. Therefore, it is hypothesized that a larger injection volume of local anaesthetic could migrate both proximal and distal within the above-described canal, spreading to additional local cutaneous nerves arising from LFCN, or even other nerves (iliohypogastric, ilioinguinal or subcostal), thereby giving rise to a greater blocked distribution area. An unwanted result of a larger injection volume is the possibility of involvement of the femoral nerve, which would result in motoric blockage of the Quadriceps muscle. It has previously been described that Iliac fascia block (injection profound to the iliaca fascia) has a great diversity in area distribution as well as blockage of the femoral nerve. By injecting the local anaesthetic directly into LFCN own canal we seek to minimize the risk of femoral nerve involvement.

Methods:

Prior to applying the nerve block, the measurement methods are tested and baseline values are registered for each leg of each participant.

The effect of a nerve block in healthy individuals can be studied by a number of validated measurement techniques. These techniques consist of mapping the affected anatomical area with temperature discrimination test (cold sensation) by using alcohol soaked gauze and pin-prick test by using a Von Frey filament, and of pain during tonic heat-stimulation of the skin (VAS tonic heat stimulation). The distribution of the sensory block is thus evaluated by high precision.

It is furthermore important to investigate whether the nerve blockade affects the femoral nerve's motorial innervation by testing m.Quadriceps' motoric function.

Course of study:

1. Baseline values are measured.
2. An orthopedic surgeon draws two hypothetical incisional lines corresponding to the posterior and to the anterior-lateral access to the hip joint on each leg of each participant. The incisional lines will be drawn with UV paint only visible under UV light. No other than the person drawing the lines and the participant will see where the lines are drawn.
3. An ultrasound guided LFCN block is then applied by a doctor with extensive experience in applying ultrasound guided blocks. Each trial participant will get two injection of Ropivacaine 0.75%. 8 ml in one leg and 16 ml in the other leg. Neither trial participants, doctors,investigator or outcome assessors will know which volume the participant receives in which leg, that is the trial is blinded.
4. After the LFCN block is applied a line called "Line A" is drawn on each leg. Line A goes from trochanter major to the femoral lateral epicondyle and is extended cranial. A line 0A is drawn perpendicular on line A at the trochanter major point. 5 cm above line 0A, is line -1A drawn up to -3A, and 5 cm below line 0A is line 1A drawn, and so forth to line 15A is reached.
5. One hour after the nerve block is applied to the right leg, the motorial and sensorial tests will be carried out on each leg, and the outcome will be registered and documented with photography. The test will be carried out on the right leg and then on the left leg in following order:

   * Maximum isometric voluntary contraction
   * Temperature discrimination test (alcohol soaked gauze)
   * Pin-prick (Von Frey filament)
   * Photo documentation
   * Drawing of the incisional lines under UV-light
   * Photo documentation
   * Measurement of the incisional lines
   * Pain stimulation test. The subjects will be monitored with blood pressure, pulse oximetry and ECG during the trial. The study extends for each participant from the introductory conversation to all testing is complete.

ELIGIBILITY:
Inclusion Criteria:

* Participant who have given their written consent after understanding the content and limitations of the study.
* ASA 1-2
* BMI ≥ 18 or ≤ 30

Exclusion Criteria:

* Participants who can not cooperate in the study.
* Participants who can not speak or understand danish.
* Allergies to the drugs used in the study.
* Alcohol abuse, by the investigators judgement.
* Drug abuse, by the investigators judgement.
* Daily use of prescription required analgesic drugs within the last four weeks.
* Consumption of over the counter analgesic drugs within the last 48 hours.
* Neuromuscular defects, former surgery or trauma to the lower extremities. (Hip to knee)
* Broken skin or wounds on the lower extremities, that could be hindering in the evaluation of the anatomical distribution of the LFCN block.
* Diabetes Mellitus.
* Pregnant women (women in the fertile age must be using safe contraception and produce a negative urine-HCG test to be able to participate in the study).
* Large tattoos in the examination area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage coverage of the incision (posterior approach) assessed by cold sensation with an alcohol swab. | 1 hour post-block
  Difference in the percentage coverage of the incision (posterior approach) between the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml, assessed by cold sensation with an alcohol swab.

SECONDARY OUTCOMES:
Difference in the percentage coverage of the incision (anterolateral approach) assessed by cold sensation with an alcohol swab. | 1 hour post-block
  Difference in the percentage coverage of the incision (anterolateral approach) between the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml, assessed by cold sensation with an alcohol swab.
Difference in the percentage coverage of the incision (posterior approach) assessed by pinprick (von frey). | 1 hour post-block
  Difference in the percentage coverage of the incision (posterior approach) between the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml, assessed by pinprick (von frey).
Difference in the percentage coverage of the incision (anterolateral approach) assessed by pinprick (von frey). | 1 hour post-block
  Difference in the percentage coverage of the incision (anterolateral approach) between the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml, assessed by pinprick (von frey).
The percentage of patients with no sensory function assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (posterior approach) on the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml.
The percentage of patients with no sensory function assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (posterior approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (posterior approach) on the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml.
The percentage of patients with no sensory function assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (anterolateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most superior part of the incision (anterolateral approach) on the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml.
The percentage of patients with no sensory function assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (anterolateral approach) | 1 hour post-block
  The percentage of patients with no sensory function (VAS = 0) assessed by Maximum pain during tonic heat stimulation test on the most inferior part of the incision (anterolateral approach) on the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml.
Estimation of the areal of the sensory loss | 1 hour post-block
  Estimation of the areal of the sensory loss (including photodocumentation) on the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml. Marked with the incisions
The difference in MVIC of the knee joint | 1 hour post-block
  The difference in MVIC (maximal voluntary isometric contraction) of the knee joint between the side given ropivacaine, 16 ml, versus the side given ropivacaine, 8 ml compared to pre-block values.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, MD, PhD, Study Chair — Naestved Hospital; Kasper H Thybo, MD, Principal Investigator — Naestved Hospital
Locations (1):
- Zealand University Hospital, Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Yes
If data is requested by an editor, it will be allowed.

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296
- [Background] Fischer HB, Simanski CJ. A procedure-specific systematic review and consensus recommendations for analgesia after total hip replacement. Anaesthesia. 2005 Dec;60(12):1189-202. doi: 10.1111/j.1365-2044.2005.04382.x. PMID 16288617
- [Background] Thybo KH, Schmidt H, Hagi-Pedersen D. Effect of lateral femoral cutaneous nerve-block on pain after total hip arthroplasty: a randomised, blinded, placebo-controlled trial. BMC Anesthesiol. 2016 Mar 23;16:21. doi: 10.1186/s12871-016-0183-4. PMID 27006014
- [Background] Thybo KH, Mathiesen O, Dahl JB, Schmidt H, Hagi-Pedersen D. Lateral femoral cutaneous nerve block after total hip arthroplasty: a randomised trial. Acta Anaesthesiol Scand. 2016 Oct;60(9):1297-305. doi: 10.1111/aas.12764. Epub 2016 Jul 18. PMID 27426231
- [Background] Doklamyai P, Agthong S, Chentanez V, Huanmanop T, Amarase C, Surunchupakorn P, Yotnuengnit P. Anatomy of the lateral femoral cutaneous nerve related to inguinal ligament, adjacent bony landmarks, and femoral artery. Clin Anat. 2008 Nov;21(8):769-74. doi: 10.1002/ca.20716. PMID 18942079
- [Background] Surucu HS, Tanyeli E, Sargon MF, Karahan ST. An anatomic study of the lateral femoral cutaneous nerve. Surg Radiol Anat. 1997;19(5):307-10. doi: 10.1007/BF01637599. PMID 9413078
- [Background] Grothaus MC, Holt M, Mekhail AO, Ebraheim NA, Yeasting RA. Lateral femoral cutaneous nerve: an anatomic study. Clin Orthop Relat Res. 2005 Aug;(437):164-8. doi: 10.1097/01.blo.0000164526.08610.97. PMID 16056045
- [Background] Dimitropoulos G, Schaepkens van Riempst J, Schertenleib P. Anatomical variation of the lateral femoral cutaneous nerve: a case report and review of the literature. J Plast Reconstr Aesthet Surg. 2011 Jul;64(7):961-2. doi: 10.1016/j.bjps.2010.11.020. Epub 2011 Jan 3. PMID 21208836
- [Background] Davies A, Crossley A, Harper M, O'Loughlin E. Lateral cutaneous femoral nerve blockade-limited skin incision coverage in hip arthroplasty. Anaesth Intensive Care. 2014 Sep;42(5):625-30. doi: 10.1177/0310057X1404200513. PMID 25233177
- [Background] Corujo A, Franco CD, Williams JM. The sensory territory of the lateral cutaneous nerve of the thigh as determined by anatomic dissections and ultrasound-guided blocks. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):561-4. doi: 10.1097/AAP.0b013e318261c8b6. PMID 22878522
- [Background] Tomaszewski KA, Popieluszko P, Henry BM, Roy J, Sanna B, Kijek MR, Walocha JA. The surgical anatomy of the lateral femoral cutaneous nerve in the inguinal region: a meta-analysis. Hernia. 2016 Oct;20(5):649-57. doi: 10.1007/s10029-016-1493-7. Epub 2016 Apr 26. PMID 27115766
- [Background] Rudin D, Manestar M, Ullrich O, Erhardt J, Grob K. The Anatomical Course of the Lateral Femoral Cutaneous Nerve with Special Attention to the Anterior Approach to the Hip Joint. J Bone Joint Surg Am. 2016 Apr 6;98(7):561-7. doi: 10.2106/JBJS.15.01022. PMID 27053584
- [Background] Hanna A. The lateral femoral cutaneous nerve canal. J Neurosurg. 2017 Mar;126(3):972-978. doi: 10.3171/2016.1.JNS152262. Epub 2016 Apr 22. PMID 27104839
- [Background] Shariat AN, Hadzic A, Xu D, Shastri U, Kwofie K, Gandhi K, McCally CM, Gratenstein K, Vandepitte C, Gadsden J, Unis D. Fascia lliaca block for analgesia after hip arthroplasty: a randomized double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2013 May-Jun;38(3):201-5. doi: 10.1097/AAP.0b013e31828a3c7c. PMID 23558369
- [Derived] Vilhelmsen F, Nersesjan M, Andersen JH, Danker JK, Broeng L, Hagi-Pedersen D, Mathiesen O, Thybo KH. Lateral femoral cutaneous nerve block with different volumes of Ropivacaine: a randomized trial in healthy volunteers. BMC Anesthesiol. 2019 Aug 28;19(1):165. doi: 10.1186/s12871-019-0833-4. PMID 31455249